CLINICAL TRIAL: NCT05233124
Title: A Randomized Controlled Trial of Dual Antiplatelet Therapy Versus Antiplatelet Monotherapy and Oral Anticoagulation in Patients With Acute Coronary Syndrome and Coronary Artery Ectasia: OVER-TIME
Brief Title: Antithrombotic Therapy in Acute Coronary Syndromes and Coronary Artery Ectasia
Acronym: OVER-TIME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Diego Araiza-Garaygordobil, Principal investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1248
Record Dates: First submitted 2022-01-14; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Ectasia
Keywords: Coronary artery ectasia; Antithrombotic therapy; Acute coronary syndrome; Coronary dilatation
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Aneurysm | interventions — Rivaroxaban; Clopidogrel; Aspirin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual antiplatelet therapy (Active Comparator): Acetyl salicylic acid, 100mg once a day + clopidogrel 75mg, once a day.
  Interventions: Drug: Acetylsalicylic acid 100mg; Drug: Clopidogrel 75 Mg Oral Tablet
- Antiplatelet monotherapy + low dose anticoagulant (Experimental): Clopidogrel 75mg + Rivaroxaban 75mg
  Interventions: Drug: Rivaroxaban 15 MG; Drug: Clopidogrel 75 Mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 15 MG — Rivaroxaban 15mg
  Other Names: Clopidogrel 75mg
  Arms: Antiplatelet monotherapy + low dose anticoagulant
Drug: Acetylsalicylic acid 100mg — Acetylsalicylic acid 100mg
  Other Names: Aspirin
  Arms: Dual antiplatelet therapy
Drug: Clopidogrel 75 Mg Oral Tablet — Clopidogrel 75mg
  Other Names: Plavix

SUMMARY:
The optimal anti-thrombotic therapy to prevent recurrent ischemic events in patients with acute coronary syndrome and coronary artery ectasia (CAE) remains unclear.

OVER-TIME is an investigator initiated, exploratory, open label, single center, randomized clinical trial comparing dual antiplatelet therapy (acetyl-salicylic acid plus a P2Y12 inhibitor) with the combination of an antiplatelet monotherapy (a P2Y12 inhibitor) plus a low dose anticoagulant (rivaroxaban, 15mg oral dose) for the prevention of recurrent ischemic events among patients with CAE. The investigators aim to enroll 60 patients with CAE and acute coronary syndromes. After recruitment, patients are randomized to (a) standard of care (dual antiplatelet regimen) or (b) the combination of antiplatelet monotherapy and low dose anticoagulant. Patients will be followed for at least 12 months. The OVER-TIME study aims to assess the efficacy of the regimen in prevention of major cardiovascular events and its security in bleeding events in acute coronary syndromes among patients with CAE.

OVER-TIME is the first randomized controlled trial to assess different antithrombotic strategies in patients with CAE and acute coronary syndrome, and its results will offer preliminary data for the prevention of major cardiovascular events and bleeding events in this group of patients.

DETAILED DESCRIPTION:
Coronary artery ectasia (CAE) is defined as a segmental or diffuse abnormal dilatation that exceeds more than 1.5 times the diameter of a normal adjacent coronary segment. The prevalence of CAE ranges from 0.3 to 4.9% and atherosclerosis is believed to be the most common etiology. According to angiographic findings, blood flow might be altered by the inappropriate dilatation in the affected arteries resulting in platelet activation and thrombus formation. Also, the presence of CAE has been related with elevated inflammatory markers and plasma soluble adhesion molecules which are an important component of vascular aneurysm formation.

Patients with MI and CAE have an increased risk of major adverse cardiovascular events (MACE) compared with those without CAE. However, it is unclear which is the optimal antithrombotic therapy for the prevention of recurrent ischemic events in patients with CAE after acute coronary syndrome (ACS)

OVER-TIME will be the first randomized controlled trial to provide insight into the safety and efficacy of different antithrombotic strategies in patients with CAE after an ACS event.

OVER- TIME is an investigator initiated, exploratory, open label, single center, randomized clinical trial comparing dual antiplatelet therapy (acetyl-salicylic acid plus a P2Y12 inhibitor) versus the combination of antiplatelet monotherapy (P2Y12 inhibitor) plus low dose anticoagulant (rivaroxaban, 15mg oral dose) for prevention of recurrent ischemic events in patients with established CAE and ACS. The trial protocol received local research and ethics committee approval and complies with the principles of the Declaration of Helsinki. Written informed consent was obtained from all patients prior to randomization.

Study patients are aged 18 or more, hospitalized with the diagnosis of ACS (NSTEMI & STEMI) undergoing coronary angiogram showing CAE in the infarction culprit artery. CAE is defined as segmental or diffuse abnormal dilatation that exceeds more than 1.5 times the diameter of a normal adjacent coronary segment. The definition of a CAE case will be based on the opinion of two independent interventional cardiologists.

The study is considered a pilot, because no randomized controlled trial has been performed to compare the efficacy of different types of antithrombotic regimens in patients with CAE after ACS. Considering a power (1-β) of 80%, an alpha level of 0.05%, accounting on the event rates of approximately 5% in patients with oral anticoagulation versus 33% in patients with dual antiplatelet therapy at 1 year of follow- up, and assuming 10% losses, the investigators calculated a sample size of 60 patients (30 per arm) for the study.

Patients are screened for the eligibility criteria during hospitalization and are randomized using 4x4 permuted blocks, after providing informed consent. Patients and treating physicians are not blinded to the allocation arm.

Patients are randomized in a 1:1 ratio to receive during 12 months a daily oral dose of DAPT (acetyl-salicylic acid 100 mg and clopidogrel 75 mg) or the combination of SAPT (clopidogrel 75 mg) and low dose of anticoagulant (rixaroxaban 15 mg). Patients will be followed for 12 months in 3 pre-specified visits (30 days, 6 months and 12 months after hospitalization). At each visit, basic clinical data will be recorded and clinical events (both ischemic and hemorrhagic, as well as safety and adverse drug events) will be actively screened.

The study has 2 co-primary endpoints, including (1) efficacy in prevention of MACE defined as the composite of cardiovascular death, non-fatal infarction, and repeated revascularization; and (2) security in major and minor bleeding, defined as a composition of major and minor bleeding events using the Bleeding Academic Research Consortium (BARC) classification.

Additionally, there are 3 secondary endpoints, including (1) the composite of net clinical benefit defined as a composite of cardiovascular death, non-fatal infarction, repeated revascularization, and major & minor bleeding events according to the BARC classification; (2) the individual components of the 2 co-primary endpoints, and (3) to compare the fibrin clot properties, by the analysis of clot lysis time and maximum turbidity, at recruitment and at 6 month of treatment.

Other clinically relevant variables such as baseline characteristics, personal history, clinical presentation, LVEF, high sensitivity cardiac troponin, NTproBNP, renal function, interventional aspects of treatment (such as stent placement, number of affected vessels, quantitative coronary angiography characterization) and other concomitant treatments will also be measured by the research staff during index event and subsequent visits.

Both the co-primary endpoints will be evaluated using the time to the occurrence of the first event. Time to the occurrence of the primary outcome and its components will be evaluated with Kaplan- Meier estimates, Log Rank Test and Cox proportional hazard models. Alternatively, analysis by "Win ratio" will be performed. For secondary outcomes, chi-squared test, T test or Wilcoxon Rank- Summation Test will be used, as appropriate.

Plasma samples will be collected from patients randomized in any group of antithrombotic therapy to analyze fibrin clots with special interest to study clot lysis time and maximum turbidity (a measure of clot density) to determine fibrin clot properties associated with clinical outcomes following CAE and ACS. This analysis may provide additional, surrogate data, as clot lysis time has been significantly associated with a higher risk of recurrent ischemic events in the long term () .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Hospitalized male or female aged >18 years.
* First event of ACS (including both, ST- Segment Elevation or Non- ST Elevation Myocardial Infarction) with high sensitivity troponin T levels exceeding 99th percentile or segmental motion abnormalities by echocardiography.
* Angiographic evidence of CAE involving the infarction culprit artery.
* Hospital length of stay >24 hours.
* Percutaneous revascularization or medical treatment according to the treating physician criteria.

Exclusion Criteria:

* Indication for temporary or permanent anticoagulation.
* Relative or absolute contraindications to receive anticoagulation.
* Chronic kidney disease (CKD) KDIGO > III or GFR <30 ml/min/1.73 m2
* Angiographic evidence of coronary aneurysms (saccular or fusiform)
* Patients undergoing coronary artery bypass graft (CABG).
* Left ventricular ejection fraction <40%.
* History of major bleeding events.
* Pregnant women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, recurrent MI and repeated revascularization | 1 year.
  Main efficacy combined outcome of cardiovascular death, recurrent MI and repeated revascularization
Composite of minor and major bleeding events. | 1 year
  Main safety combined outcome of minor and major events, measured by BARC scale.

SECONDARY OUTCOMES:
Net clinical benefit composite endpoint, including cardiovascular death, recurrent MI, repeated revascularization and minor/major bleeding | 1 year
  Composite of cardiovascular death, recurrent MI, repeated revascularization and minor/major bleeding
Clot lysis time by turbidimetry | 6 months
  Time (in seconds) taken for turbidity to drop by 50% from maximum as a measure of lysis potential

CONTACTS AND LOCATIONS:
Overall Officials: Diego Araiza Garaygordobil, MD, MSc, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; Alexandra Arias Mendoza, MD, Study Director — Instituto Nacional de Cardiología Ignacio Chávez
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cardiologia, Mexico City
  - Instituto Nacional de Cardiología "Ignacio Chavez", Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Araiza-Garaygordobil D, Gopar-Nieto R, Sierra-Lara Martinez JD, Mullasari AS, Belderrain-Morales N, Najera-Rojas NA, Diaz-Herrera BA, Sarabia-Chao V, Alfaro-Ponce DL, Briseno-De la Cruz JL, Ruiz-Beltran M, Martinez-Rios MA, Pina-Reyna Y, Latapi-Ruiz Esparza X, Grimaldo-Gomez FA, Cortina-De la Rosa E, Romero-Arroyo MO, Sierra-Gonzalez de Cossio A, Gonzalez-Pacheco H, Arias-Mendoza A. A randomized trial of antithrombotic therapy in patients with acute coronary syndrome and coronary ectasia. Am Heart J. 2025 Mar;281:103-111. doi: 10.1016/j.ahj.2024.11.012. Epub 2024 Nov 29. PMID 39615618
- [Derived] Araiza-Garaygordobil D, Gopar-Nieto R, Sierra-Lara Martinez D, Belderrain-Morales N, Sarabia-Chao V, Alfaro-Ponce DL, Ontiveros-Mercado H, Mendoza-Garcia S, Altamirano-Castillo A, Martinez-Amezcua P, Cabello-Lopez A, Briseno-De la Cruz JL, Ruiz-Beltran M, Martinez-Rios MA, Pina-Reyna Y, Gonzalez-Pacheco H, Arias-Mendoza A. Dual Antiplatelet Therapy Versus Antiplatelet Monotherapy Plus Oral Anticoagulation in Patients with Acute Coronary Syndrome and Coronary Artery Ectasia: Design and Rationale of OVER-TIME Randomized Clinical Trial. High Blood Press Cardiovasc Prev. 2022 Sep;29(5):463-468. doi: 10.1007/s40292-022-00535-4. Epub 2022 Jul 29. PMID 35904750